CLINICAL TRIAL: NCT06414408
Title: Randomized Directly Observed Therapy Study to Interpret Clinical Trials of Doxy-PEP
Acronym: DOT-Doxy-PEP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AI186641; R01AI186641 (NIH)
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Sexually Transmitted Diseases, Bacterial
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of 4 doxycycline dosing patterns (daily, 3x weekly, weekly, every other week) and then will crossover to an alternate pattern once during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Daily Dosing (Active Comparator): Participants will be randomized to take once daily doxycycline 200mg for six weeks.
  Interventions: Drug: Doxycycline Pill
- Three-times Weekly Dosing (Active Comparator): Participants will be randomized to take one doxycycline 200mg dose three times a week (Monday, Wednesday, and Friday) for six weeks.
  Interventions: Drug: Doxycycline Pill
- Weekly Dosing (Active Comparator): Participants will be randomized to take one doxycycline 200mg dose once week.
  Interventions: Drug: Doxycycline Pill
- Every Other Week Dosing (Active Comparator): Participants will be randomized to take one doxycycline 200mg dose every other week.
  Interventions: Drug: Doxycycline Pill

INTERVENTIONS:
Drug: Doxycycline Pill — 200mg Dose

SUMMARY:
Rates of bacterial sexually transmitted infections (STIs) are rising globally, demanding innovative interventions beyond the scope of current efforts to prevent STIs. The United States Doxycycline Post-exposure Prophylaxis (DoxyPEP) Study has demonstrated the efficacy of doxycycline post-exposure prophylaxis (PEP) among men who have sex with men and transgender women; but puzzlingly, doxycycline PEP was found ineffective in cisgender women in the Kenyan doxycycline Post-Exposure Prophylaxis (dPEP) study, with preliminary data suggesting the low medication adherence may explain the null result. By study end, the investigators will have developed adherence measurement methods for doxycycline in hair, blood, and urine, and will use these techniques to help interpret the Kenyan dPEP study, and to examine the relative performance of these methods within the United States DoxyPEP trial, establishing adherence metrics for current and future rollout studies of doxycycline post-exposure prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* not currently at risk of a sexually transmitted infection and willing to use other methods, such as condoms, for STI prevention;
* if diagnosed with an STI in the past two years and/or a partner was diagnosed with an STI in the past year, is willing to use condoms for STI prevention;
* willing to provide hair, blood, and urine samples;
* not currently enrolled in other STI prevention studies;
* able to speak English
* transgender women participants should be currently using estrogen gender affirming hormone therapy with blood estrogen levels demonstrating consistent use
* transgender men participants should be currently using testosterone gender affirming hormone therapy with blood testosterone levels demonstrating consistent use
* able to provide a hair sample of ~50-100 strands of hair that are non-gray, not bleached, and at least 1cm in length
* willing to NOT shave hair or have a very short haircut or apply bleach for the duration of the study
* has suitable venous access for consecutive blood draws

Exclusion Criteria:

* any health condition that may interfere with participation or the ability to provide informed consent, including any debilitating or life-threatening conditions;
* pregnancy or plans to become pregnant;
* liver cirrhosis or fulminant liver disease;
* known hypersensitivity reaction to doxycycline.
* detectable doxycycline in hair at enrollment.
* unable to provide a hair sample of ~50-100 strands of hair that are non-gray, not bleached, and at least 1cm in length
* does not have suitable venous access for consecutive blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Hair Doxycycline Concentration | 4 weeks
  Doxycycline concentrations will be measured using liquid chromatography tandem mass spectrometry within hair samples for each of the four dosing patterns within an intensive washout pharmacokinetic phase following initial dosing.
Plasma Doxycycline Concentration | 4 weeks
  Doxycycline concentrations will be measured using liquid chromatography tandem mass spectrometry within plasma samples for each of the four dosing patterns within an intensive washout pharmacokinetic phase following initial dosing.
Urine Doxycycline Concentration | 4 weeks
  Doxycycline concentrations will be measured using liquid chromatography tandem mass spectrometry within urine samples for each of the four dosing patterns within an intensive washout pharmacokinetic phase following initial dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Spinelli, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco/San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No